CLINICAL TRIAL: NCT04647253
Title: AGENT IDE: A Prospective, Randomized (2:1), Multicenter Trial to Assess the Safety and Effectiveness of the AgentTM Paclitaxel Coated PTCA Balloon Catheter for the Treatment of Subjects With In-Stent Restenosis (ISR)
Brief Title: A Clinical Trial to Assess the Agent Paclitaxel Coated PTCA Balloon Catheter for the Treatment of Subjects With In-Stent Restenosis (ISR)
Acronym: AGENT IDE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2358
Record Dates: First submitted 2020-11-23; First posted 2020-11-30 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: In-Stent Restenosis
Keywords: Drug coated balloon

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized (2:1), Multicenter Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AGENT DCB (Experimental): Agent DCB is a Monorail Percutaneous Transluminal Coronary Angioplasty (PTCA) balloon catheter with a semi-compliant balloon coated with a formulation of paclitaxel (drug) and an excipient, Acetyl-Tri-n-butyl citrate (ATBC). The balloon catheter platform is based on the commercially available BSC Emerge™ PTCA balloon catheter system (K130391).
  Interventions: Device: AGENT DCB
- Commercially available, PTCA Dilation Catheter (Active Comparator)
  Interventions: Device: PTCA balloon catheter

INTERVENTIONS:
Device: AGENT DCB — Drug coated PTCA balloon catheter
  Arms: AGENT DCB
Device: PTCA balloon catheter — PTCA balloon catheter
  Arms: Commercially available, PTCA Dilation Catheter

SUMMARY:
AGENT IDE is a Prospective, Randomized (2:1), Multicenter Trial. The purpose of this study is to assess the safety and effectiveness of the Agent Paclitaxel Coated PTCA Balloon Catheter compared to balloon angioplasty (POBA) in patients with in-stent restenosis (ISR) of a previously treated lesion of up to 26 mm in length (by visual estimate) in a native coronary artery 2.0 mm to 4.0 mm in diameter.

ELIGIBILITY:
Clinical Inclusion Criteria

* Subject must be at least 18 years of age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures, and provides written informed consent before any trial-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI)
* Subject is willing to comply with all protocol-required follow-up evaluation
* Women of child-bearing potential must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure

Angiographic Inclusion Criteria (visual estimate)

* In-stent restenosis in a lesion previously treated with either a drug-eluting stent or bare metal stent, located in a native coronary artery with a visually estimated reference vessel diameter (RVD) > 2.0 mm and ≤ 4.0 mm.
* Target lesion length must be < 26 mm (by visual estimate) and must be covered by only one balloon.
* Target lesion must have visually estimated stenosis > 50% and < 100% in symptomatic patients (>70% and <100% in asymptomatic patients) prior to lesion pre-dilation.
* Target lesion must be successfully pre-dilated.

  o Note: Successful predilation/pretreatment refers to dilation with a balloon catheter of appropriate length and diameter, or pretreatment with directional or rotational coronary atherectomy, laser or cutting/scoring balloon with no greater than 50% residual stenosis and no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C. Thrombolysis in Myocardial Infarction (TIMI) grade flow in the target lesion must be >2
* If a non-target lesion is treated, it must be treated first and must be deemed a success.

  * Note: Successful treatment of a non-target lesion is defined as a residual stenosis of ≤ 30% in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of prolonged chest pain or ECG changes consistent with MI.

Clinical Exclusion Criteria

* Subject has other serious medical illness (e.g. cancer, congestive heart failure) that may reduce life expectancy to less than 24 months.
* Subject has current problems with substance abuse (e.g. alcohol, cocaine, heroin, etc.).
* Subject has planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* Subject is participating in another investigational drug or device clinical study that has not reached its primary endpoint.
* Subject intends to participate in another investigational drug or device clinical study within 12 months after the index procedure.
* Woman who is pregnant or nursing. (A pregnancy test must be performed within 7 days prior to the index procedure, except for women who definitely do not have child-bearing potential.)
* Left ventricular ejection fraction known to be < 25%.
* Subject had PCI or other coronary interventions within the last 30 days.
* Planned PCI or CABG after the index procedure.
* STEMI or QWMI <72h prior to the index procedure.
* Cardiogenic shock (SBP < 80 mmHg requiring inotropes, IABP or fluid support).
* Known allergies against paclitaxel or other components of the used medical devices.
* Known hypersensitivity or contraindication for contrast dye that in the opinion of the investigator cannot be adequately pre-medicated.
* Intolerance to antiplatelet drugs, anticoagulants required for procedure.
* Platelet count < 100k/mm3 (risk of bleeding) or > 700k/mm3.
* Subject with renal insufficiency (creatinine ≥2.0 mg/dl) or failure (dialysis dependent).
* Subject has suspected or proven COVID-19 at present or within the past 4 weeks with resolution of symptoms.

Angiographic Exclusion Criteria (visual estimate)

* Target lesion is located within a bifurcation with planned treatment of side branch vessel.
* Target lesion is located within a saphenous vein or arterial graft.
* Thrombus present in the target vessel
* > 50% stenosis of an additional lesion proximal or clinically significant distal (>2.0mm RVD) to the target lesion.
* Patient with unprotected left main coronary artery disease. (>50% diameter stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yeh, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (40):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Carondelet Medical Group St. Mary's Hospital, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - St. Anthony Hospital, Lakewood, Colorado
  - South Denver Cardiology, Littleton, Colorado
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Evanston Hospital, Evanston, Illinois
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Bergan Cardiology, Omaha, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Wake Medical Center, Raleigh, North Carolina
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UPMC Pinnacle Health, Wormleysburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Methodist North Hospital, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Yeh RW, Bachinsky W, Stoler R, Bateman C, Tremmel JA, Abbott JD, Dohad S, Batchelor W, Underwood P, Allocco DJ, Kirtane AJ. Rationale and design of a randomized study comparing the agent drug coated balloon to plain old balloon angioplasty in patients with In-stent restenosis. Am Heart J. 2021 Nov;241:101-107. doi: 10.1016/j.ahj.2021.07.008. Epub 2021 Jul 24. PMID 34314727
- [Result] Yeh RW, Shlofmitz R, Moses J, Bachinsky W, Dohad S, Rudick S, Stoler R, Jefferson BK, Nicholson W, Altman J, Bateman C, Krishnaswamy A, Grantham JA, Zidar FJ, Marso SP, Tremmel JA, Grines C, Ahmed MI, Latib A, Tehrani B, Abbott JD, Batchelor W, Underwood P, Allocco DJ, Kirtane AJ; AGENT IDE Investigators. Paclitaxel-Coated Balloon vs Uncoated Balloon for Coronary In-Stent Restenosis: The AGENT IDE Randomized Clinical Trial. JAMA. 2024 Mar 26;331(12):1015-1024. doi: 10.1001/jama.2024.1361. PMID 38460161
- [Derived] Jamil Y, Kirtane A, Yeh RW, Shlofmitz R, Moses J, Bachinsky W, Dohad S, Rudick S, Stoler R, Jefferson BK, Nicholson W, Altman J, Krishnaswamy A, Alaswad K, Kimmelstiel C, Reitman A, Cavalcante R, Tehrani BN, Batchelor WB. Paclitaxel-Coated Balloon for Treating In-Stent Restenosis in Racial and Ethnic Minority Patients: A Subanalysis From the AGENT IDE Trial. J Am Heart Assoc. 2026 Jan 19:e043053. doi: 10.1161/JAHA.125.043053. Online ahead of print. PMID 41553096
- [Derived] Wen J, Dohad S, Shlofmitz R, Moses J, Bachinsky W, Rudick S, Stoler R, Jefferson BK, Nicholson W, Altman J, Neupane S, Croce K, Shunk K, Taylor A, Saybolt MD, Diaz C, Cavalcante R, Yeh RW, Kirtane AJ. Paclitaxel-Coated Balloon for the Treatment of Small Vessel In-Stent Restenosis: A Subgroup Analysis of the AGENT IDE Randomized Trial. JACC Cardiovasc Interv. 2025 Nov 24;18(22):2701-2710. doi: 10.1016/j.jcin.2025.09.032. PMID 41297981
- [Derived] Kirtane AJ, Shlofmitz R, Moses J, Bachinsky W, Dohad S, Rudick S, Stoler R, Jefferson BK, Nicholson W, Altman J, Bateman C, Krishnaswamy A, Grantham JA, Zidar FJ, Tremmel JA, Grines C, Ahmed MI, Latib A, Tehrani B, Abbott JD, Batchelor W, Cavalcante R, Yeh RW. Paclitaxel-Coated Balloon for the Treatment of Multilayer In-Stent Restenosis: AGENT IDE Subgroup Analysis. J Am Coll Cardiol. 2025 Aug 19;86(7):502-511. doi: 10.1016/j.jacc.2025.05.062. PMID 40803784

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGENT DCB | Commercially Available, PTCA Dilation Catheter
Started | 406 | 194
Completed (12-Month clinical follow-up performed, with visit window of 365 +/- 30 days) | 373 | 176
Not Completed | 33 | 18
Not completed — Death ≤ 365 Days | 16 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Missed 12-Month Visit | 9 | 7
Not completed — Death > 365 days and ≤ 395 days with no 12-month clinical follow-up performed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGENT DCB | Commercially Available, PTCA Dilation Catheter | Total
Number analyzed (Participants) | 406 | 194 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.42 (9.79) | 67.90 (9.68) | 68.25 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 53 | 157
  Male | 302 | 141 | 443
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnicity were combined into a single question in the electronic database. Sites were instructed to check all that apply. This could have included only checking 'Hispanic or Latino'. Therefore, the sum of the race and ethnicity categories may not equal the number of participants analyzed in each arm/group.
  Participants
    American Indian or Alaska native | 0 | 1 | 1
    Asian | 9 | 6 | 15
    Black, of African heritage | 32 | 10 | 42
    Caucasian | 304 | 148 | 452
    Hispanic or Latino | 26 | 9 | 35
    Native Hawaiian or other Pacific Islander | 1 | 1 | 2
    Other | 16 | 3 | 19
    Not Disclosed | 23 | 18 | 41
Region of Enrollment [Number; unit: participants]
  United States | 406 | 194 | 600
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: Number analyzed excludes subjects listed as unknown
  kg/m2
    number analyzed (Participants) | 396 | 191 | 587
    (all) | 30.01 (5.53) | 30.10 (5.85) | 30.04 (5.64)
Current Diabetes Mellitus [Count of Participants; unit: Participants] — Population: Number analyzed excludes subjects listed as unknown
  Participants
    number analyzed (Participants) | 404 | 194 | 598
    (all) | 206 | 97 | 303
History of Myocardial Infarction [Count of Participants; unit: Participants] — Population: Number analyzed excludes subjects listed as unknown
  Participants
    number analyzed (Participants) | 398 | 190 | 588
    (all) | 198 | 95 | 293
Stent Layer in Target Lesion [Count of Participants; unit: Participants]
  Single Layer | 230 | 112 | 342
  Multiple Layers | 176 | 82 | 258

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Lesion Failure
Description: The primary endpoint is the 12-month Target Lesion Failure (TLF) rate, defined as any ischemia-driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death
Time Frame: 12-month
Population: The number of participants analyzed excludes subjects with insufficient follow up (i.e. subjects were followed less than 335 days post-procedure) and without experiencing 12-month TLF
Measure: Count of Participants; unit: Participants
Arm/Group | AGENT DCB | Commercially Available, PTCA Dilation Catheter
Number analyzed (Participants) | 390 | 186
Participants | 71 | 54
Statistical Analysis 1: Comparison: AGENT DCB vs Commercially Available, PTCA Dilation Catheter; Test type: Superiority; p = 0.0025, z-test with unpooled variance — a priori threshold for statistical significance was 0.025; Rate difference between treatment groups = -10.8, 95% CI 2-sided [-18.4 to -3.3]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 395 days post procedure. Serious and Other Adverse Events were monitored up to 365 days post procedure.
Description: Adverse events were assessed at each follow-up visit (30 days, 6 months, and 12 months)
Arm/Group | AGENT DCB | Commercially Available, PTCA Dilation Catheter
All-Cause Mortality (participants affected / at risk) | 17/406 | 8/194
Serious Adverse Events (participants affected / at risk) | 226/406 | 113/194
Other Adverse Events (participants affected / at risk) | 79/406 | 50/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGENT DCB (N=406) | Commercially Available, PTCA Dilation Catheter (N=194)
Angina unstable (Cardiac disorders) | 35 (43) | 25 (36)
Angina pectoris (Cardiac disorders) | 40 (43) | 23 (28)
Acute myocardial infarction (Cardiac disorders) | 21 (25) | 14 (16)
Coronary artery disease (Cardiac disorders) | 21 (21) | 11 (12)
Atrial fibrillation (Cardiac disorders) | 14 (16) | 5 (5)
Cardiac failure (Cardiac disorders) | 10 (17) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 7 (8) | 8 (10)
Myocardial infarction (Cardiac disorders) | 7 (7) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 4 (4)
Left ventricular failure (Cardiac disorders) | 3 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block right (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery perforation (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 5 (5)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Appendicitis (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Purulence (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 11 (11) | 5 (5)
Chest pain (General disorders) | 5 (5) | 3 (4)
Vascular stent stenosis (General disorders) | 5 (5) | 3 (3)
Catheter site haematoma (General disorders) | 3 (3) | 1 (1)
Catheter site haemorrhage (General disorders) | 2 (2) | 1 (1)
Death of unknown cause (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Medical device site thrombosis (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Stenosis (General disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Optic perineuritis (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 8 (8) | 3 (3)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)
Aortic stenosis (Vascular disorders) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 3 (3)
Haemodynamic instability (Vascular disorders) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Plaque shift (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Starvation ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 10 (12) | 3 (3)
Urinary retention (Renal and urinary disorders) | 5 (5) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 3 (3) | 2 (2)
Acid base balance abnormal (Investigations) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0)
Pulse absent (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia stage 3 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (4) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast conserving surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Device lead damage (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGENT DCB (N=406) | Commercially Available, PTCA Dilation Catheter (N=194)
Angina pectoris (Cardiac disorders) | 40 (42) | 20 (21)
Covid-19 (Infections and infestations) | 34 (37) | 17 (19)
Non-cardiac chest pain (General disorders) | 10 (11) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT04647253/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04647253/SAP_001.pdf